CLINICAL TRIAL: NCT02996162
Title: The Natural Course of Hypercapnia and Its Association With Long-term Respiratory Morbidities in Premature Infants With Chronic Lung Disease
Brief Title: Hypercapnia and Its Association With Long-term Respiratory Morbidities in Premature Infants With Chronic Lung Disease
Status: Withdrawn | Type: Observational
Why Stopped: The research never began; the PI has chosen to no longer pursue this project.
Sponsor: Boston Children's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Kristen Leeman, MD, Boston Children's Hospital
Other Study IDs: IRB-P00019957
Record Dates: First submitted 2016-08-30; First posted 2016-12-19 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; Chronic Lung Disease; Prematurity
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Massimo Root Monitoring System — The Masimo Root system is a patient monitoring and connectivity platform; Root displays patient monitoring information from the connected modules. This will be used as a non-invasive way to determine infants' pCO2. The equipment will be used in the inpatient portion of the study up to twice weekly for 5 minutes to obtain approximately 150 end tidal CO2 values and recorded over time for each infant. In the outpatient portion, it will be used in each clinic visit in a similar fashion.
  Other Names: Masimo Root Monitoring System and Accessories
Device: ISA-Infrared Sidestream Gas Analyzer — The ISA-Infrared Sidestream Gas Analyzer displays end-tidal carbon dioxide waveforms and measurements and trends of end tidal CO2. This will be used as a non-invasive way to determine infants' pCO2. The equipment will be used in the inpatient portion of the study up to twice weekly for 5 minutes to obtain approximately 150 end tidal CO2 values and recorded over time for each infant. In the outpatient portion, it will be used in each clinic visit in a similar fashion.
  Other Names: Infrared Sidestreamn gas Analyzer (ISA); Multigas Monitor

SUMMARY:
This is a prospective, longitudinal observational study to provide data regarding the natural course of hypercapnia in premature infants with bronchopulmonary dysplasia using both available blood pCO2 and measured capnography, as well as relate the degree and trend of hypercapnia to later respiratory outcomes.

DETAILED DESCRIPTION:
Data collection will begin once an infant no longer requires mechanical ventilation, CPAP, and HFNC, up to twice per week while in the NICU. Investigators will obtain up to twenty minutes of end-tidal capnography data, using Masimo ISA modules with continuous CO2 display. Five minutes of good quality data, at approximately 30 breaths per minutes, should provide approximately 150 data points. After filtering for artifact, the mean and range of end tidal CO2 will be recorded during this interval. These recordings will be started after a feed for infants receiving enteral feeds. The capnography cannula will be placed by the bedside nurse or respiratory therapist at the conclusion of a feed and removed no later than the next feed. If data is unable to be obtained, investigators will attempt to collect it at the next regularly scheduled interval.

Available blood gases with pCO2 will also be recorded during the NICU hospitalization.

After discharge, consented subjects who are followed in the BCH outpatient pulmonary clinic will have capnography recorded at every clinic visit for a period of up to twenty minutes, and mean and range of end-tidal CO2 will be recorded after filtering for artifact. Available blood gases with pCO2 during pulmonary visits will be recorded; blood gases during sick encounters (i.e. emergency room) will be excluded. From available electronic medical record (EMR) and clinic note data, investigators will also record duration of time on respiratory support including positive pressure ventilation and nasal cannula oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Potential eligible patients will be identified in the first 3-14 days of life at Beth Israel Deaconess Hospital (BIDMC) NICU who have a birth gestational age <=32 0/7 weeks and current or previous requirement for positive pressure (ventilation or continuous positive airway pressure (CPAP).

Exclusion Criteria:

1. death prior to discharge from the NICU,
2. chronic lung disease secondary to pulmonary conditions other than bronchopulmonary dysplasia and
3. other underlying identified genetic syndromes.

Ages: 3 Days to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants with chronic lung disease of prematurity or bronchopulmonary dysplasia
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-05-06 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Respiratory symptoms and complications | One year
  Primary outcome will be respiratory symptoms at one year. Respiratory symptoms will be measured by a parent-reported respiratory symptom score obtained via questionnaire.

SECONDARY OUTCOMES:
Respiratory support | One year
  Secondary outcomes will include respiratory support, including duration of need for positive pressure ventilation (number of days), duration of need for supplemental oxygen (number of days), and use of respiratory related medications (yes or no response as to whether used and percentage of use).
Respiratory complications | One year
  Secondary outcome will be respiratory complications at one year. Complications will include death from respiratory cause (number of deaths), readmission for respiratory illness (number of readmissions), ICU admission (number of admissions), need for reintubation or positive pressure ventilation (number of events).
Non-respiratory complications | One year
  Secondary outcomes will include non-respiratory complications such as aspiration requiring limitation of oral feeding (percentage).

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Leeman, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No